CLINICAL TRIAL: NCT04784390
Title: A 16 Week Randomized, Single-masked, Multicenter Proof of Concept Study of Binocular Videogames Versus Patching for Amblyopia in Children 4-7 Years of Age With an Open-label Substudy of Binocular Videogames in Children 8-12 Years of Age
Brief Title: Proof of Concept Study of Binocular Videogames Versus Patching for Amblyopia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated based upon the competitive landscape and strategic fit.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDDO001F12201
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Amblyopia
Keywords: DDO001; amblyopia; binocular video games; patching; eye disorder; lazy eye; unable to focus in one eye; eye muscle disorder; wandering eye; abnormal vision development
MeSH Terms: conditions — Amblyopia; Eye Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Part A: Single-masked by outcome assessor only
  Part B: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Patching (Active Comparator): Patching of the sound eye (fellow eye) - patients will have their sound eye (fellow eye) patched 2 hours per day 7 days a week for 16 weeks.
  Interventions: Device: Patching of the sound eye
- Binocular video games (Experimental): Binocular video games - patients will play 1 hour of binocular video game of choice (Dig Rush and/or Monster Burner) a day 7 days a week for 8 to 12 weeks.
  Interventions: Device: Binocular video games

INTERVENTIONS:
Device: Binocular video games — Patients will play 1 hour of binocular video game of choice (Dig Rush and/or Monster Burner) a day 7 days a week for 8 to 12 weeks.
  Arms: Binocular video games
Device: Patching of the sound eye — Patients will have their sound eye (fellow eye) patched 2 hours per day 7 days a week for 16 weeks.
  Arms: Patching

SUMMARY:
The purpose of this PoC study was to evaluate the potential therapeutic efficacy of binocular video games played on a tablet and to compare the efficacy of binocular video games versus patching in amblyopic patients 4 to 7 years old (Part A) as well as to gain experience with binocular video games in older children population of 8 to12 years old (Part B).

Part A and Part B was designed to provide long term data on durability of binocular video games treatment.

The study consisted of two parts, Part A: randomized, single masked PoC study in children 4 to 7 years old at Screening, and Part B: open-label substudy in children 8 to 12 year old at Screening.

DETAILED DESCRIPTION:
The clinical investigation consisted of 2 parts:

* Part A: a single-masked, randomized clinical investigation in subjects 4 to 7 years of age.
* Part B: an open-label, non-randomized sub-investigation in subjects 8 to 12 years of age.

Part A was a 16-week, prospective, randomized, single-masked, multicenter, controlled, 2 arm, parallel-group clinical investigation in subjects 4 to 7 years of age with amblyopia. Subjects were randomly assigned in a 1:1 ratio to either binocular videogame treatment for 8 to 12 weeks or patching treatment for 16 weeks. Randomization was stratified by severity of amblyopia in eligible subjects (moderate amblyopia with best-corrected visual acuity (BCVA) of the amblyopic eye of 20/100 or better, or severe amblyopia with BCVA of the amblyopic eye worse than 20/100).

Part B was a 16-week, open-label, single arm sub investigation in subjects 8 to 12 years of age with amblyopia, in which selected sites could participate. Subjects received binocular videogame treatment for 8 weeks, followed by 8 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be signed by the parent(s) or legal guardian(s) prior to participation in the study.
2. Male or female children 4 to 7 years old at Screening (Part A) or 8 to 12 years old at Screening (Part B).
3. Diagnosis of amblyopia due to strabismus, anisometropia, or both.
4. Best corrected visual acuity (BCVA) of amblyopic eye (study eye) between 0.3 to 1.0 Logarithm of the Minimum Angle of Resolution (logMAR) (20/40 to 20/200 Snellen inclusive, 33 to 72 ETDRS letters inclusive) at Screening and Baseline.
5. BCVA of the sound eye (fellow eye) 0.1 logMAR (20/25 Snellen, 80 Early Treatment Diabetic Retinopathy Study (ETDRS) letters) or better in children 5 years of age and older or 0.2 logMAR (20/30 Snellen, 75 ETDRS letters) or better in children 4 years of age at Screening and Baseline.
6. Interocular difference of BCVA at least 0.3 logMAR (≥3 lines; ETDRS≥15 letters) at Baseline.
7. Patient is able to play the binocular game (Dig Rush and Monster Burner) on at least level 3 on the study tablet under binocular conditions (with red-green glasses).

Exclusion Criteria:

1. Treatment for amblyopia with patching, Bangerter filter, vision therapy, or binocular treatment in the past 1 week prior to Screening, or atropine in the past 4 weeks prior to Screening.
2. Treatment for amblyopia with patching, Bangerter filter, vision therapy, binocular treatment or atropine for more than 1 year prior to screening cumulatively.
3. Myopia ≥ -6.00D spheric equivalent in either eye at Screening or Baseline.
4. Prior amblyopia treatment (patching, Bangerter filter, vision therapy, binocular treatment or atropine) for more than a year prior to screening cumulatively.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Change in best corrected visual acuity (BCVA) in the amblyopic eye. | from Baseline to Week 8
  Part A: Best corrected visual acuity (BCVA) in the amblyopic eye will be measured via mixed model repeated measures (MMRM).

SECONDARY OUTCOMES:
Attain BCVA of 0.1 logMAR or better in the amblyopic eye | at Week 4, Week 8, Week 12, and Week 16.
  Part A: Best corrected visual acuity (BCVA) in the amblyopic eye will be measured via mixed model repeated measures (MMRM).
Change in stereoacuity or binocular video game relative to patching. | from Baseline to Week 4, Week 8, Week 12, and Week 16.
  Part A: Stereoacuity will be assessed at near using Randot Preschool Stereoacuity Test (Stereo Optical, Inc.).
  The test is performed using 3 stereotest booklets while wearing 3D glasses. In short, in each test booklet, the left-hand page shows two-dimensional black-and-white silhouettes of two sets (panels) of four test shapes. The right-hand page contains two sets of four random-dot patterns in different sequences that are on the left-hand page. In each set of random-dot patterns, one contains no test shape, while the remaining contains test shapes. The child must correctly identify at least two of the three test shapes at each disparity level.
Attain a 2-line or better improvement in BCVA in the amblyopic eye | at Week 4, Week 8, Week 12, and Week 16.
  Part A: Best corrected visual acuity (BCVA) in the amblyopic eye will be measured via mixed model repeated measures (MMRM).
Change in BCVA in the amblyopic eye | from Baseline to Week 4, Week 12, and Week 16.
  Part A: Best corrected visual acuity (BCVA) in the amblyopic eye will be measured via mixed model repeated measures (MMRM).
Frequency of treatment-emergent Adverse Events | from Baseline to week 16
  Part A and B: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical study subject, user or other person, after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of the study device, i.e., videogame system (tablet, software, 3D glasses) or patch.
Time played as recorded in the diary | from Baseline to week 12
  Part A: To assess compliance with treatment
Time patched as recorded in the diary | from Baseline to week 16
  Part A: To assess compliance with treatment
Time played as recorded in the video game system | from Baseline to week 12
  Parts A and B: To assess compliance with treatment
Percentage of participants who complete at least 75% of prescribed game play | from Baseline to Week 12
  Parts A and B: To assess compliance with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (5):
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Maitland, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Frederick, Maryland
  - Novartis Investigative Site, Las Vegas, Nevada
- Novartis Investigative Site, North Ryde, New South Wales, Australia
- Canada (2):
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CDDO001F12201 from the Novartis Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18045